CLINICAL TRIAL: NCT07263165
Title: Effect of Adding Dexmedetomidine as Adjuvant to Bupivacaine in Ultrasound Guided External Oblique Intercostal Plane Block in Upper Abdominal Cancer Surgery. A Prospective Randomized Clinical Trial
Brief Title: Dexmedetomidine as an Adjuvant to Bupivacaine for Ultrasound-Guided External Oblique Intercostal Block
Acronym: Dexmedetomidin
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ibrahem Shaker, Anesthesia Resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: External Ob. intercostal block
Record Dates: First submitted 2025-11-16; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: Opioid Consumption, Postoperative
Keywords: dexmedetomidine; external oblique intercostal block
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine + Bupivacaine (Experimental): Participants will receive an ultrasound-guided external oblique intercostal plane block using 20 mL of 0.25% bupivacaine combined with dexmedetomidine (0.5 µg/kg) administered as a single-shot injection.
  Interventions: Drug: Dexmedetomidine
- Bupivicaine (Active Comparator): Participants will receive an ultrasound-guided external oblique intercostal plane block using 20 mL of 0.25% bupivacaine administered as a single-shot injection without any adjuvant.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine as Adjuvant toBupivacaine in Ultrasound Guided ExternalOblique Intercostal Plane Block

SUMMARY:
Effect of Adding Dexmedetomidine as Adjuvant toBupivacaine in Ultrasound Guided ExternalOblique Intercostal Plane Block in UpperAbdominal Cancer Surgery.

DETAILED DESCRIPTION:
Effect of Adding Dexmedetomidine as Adjuvant toBupivacaine in Ultrasound Guided ExternalOblique Intercostal Plane Block in UpperAbdominal Cancer Surgery. A prospectiverandomized clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 years scheduled for elective upper abdominal cancer surgery (e.g., gastrectomy, hepatectomy, pancreatectomy).
* American Society of Anesthesiologists (ASA) physical status I-III.
* Body mass index (BMI) between 18-35 kg/m².

Exclusion Criteria:

* Patient refusal.
* Allergy to local anesthetics or dexmedetomidine.
* Coagulopathy (INR >1.5, platelet count <100,000/mm³).
* Infection at the injection site.
* Severe cardiopulmonary, renal, or hepatic dysfunction.
* Chronic opioid use (>30 mg morphine equivalents daily for >3 months).
* Pregnancy or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Total Postoperative Opioid Consumption (mg of morphine equivalents) | 24 hours postoperative.
  To evaluate the effect of adding dexmedetomidine to bupivacaine on total opioid consumption within the first 24 hours after upper abdominal cancer surgery.

SECONDARY OUTCOMES:
Postoperative Pain Intensity Using the Visual Analog Scale (VAS 0-10) | 2, 4, 6, 12, 18, and 24 hours postoperative.
  Pain scores will be assessed at rest and during movement using the Visual Analog Scale (0 = no pain, 10 = worst pain). Higher scores indicate worse pain.
Time to First Request for Rescue Analgesia. | 24 hour postoperative
  Time from block performance until first request for analgesia.
Number of Participants with Adverse Effects | first 2 hours postoperative.
  Incidence of nausea, vomiting, hypotension, and bradycardia.
patient satisfaction score | 1 hour postoperative
  Patient satisfaction regarding pain control (0 = completely dissatisfied, 10 = fully satisfied). Higher scores indicate better satisfaction.
Block-related complications. | intraoperative and 24 postoperative
  Incidence of hematoma, infection, or local anesthetic systemic toxicity (LAST).